CLINICAL TRIAL: NCT01466400
Title: Fermentation Rate of Infant Formula
Status: Completed | Type: Observational
Sponsor: Father Flanagan's Boys' Home (Other)
Collaborators: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-18-F
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: health benefits of infant formula

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- infants two to six months of age

SUMMARY:
It is hypothesized that there will be no difference in the breath hydrogen excretion between the 2 different prebiotic formulas.

DETAILED DESCRIPTION:
This pilot study is looking at how a formula with one of two different prebiotic blends may alter the hydrogen level in an infant's exhalations in the hours after feeding. Higher levels for a longer period may signal higher levels of short chain fatty acids and bifidobacteria, both beneficial for gastrointestinal health. The higher levels may be the result of the formula undergoing a slower digestion, producing more fermentation.

The study will compare a formula, similar to one currently on the market, with added prebiotics using a special breathing mask designed to be held to the infant's mouth and nose long enough to capture the infant's exhaled breath which will then be tested for Hydrogen content.

ELIGIBILITY:
Inclusion Criteria:

* 2-6 months of age,
* healthy,receiving standard cow-milk based infant formula weight,
* greater than 5th percentile

Exclusion Criteria:

* on no antibiotics,
* breastfed,
* on solid foods

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy infants.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Hydrogen content of breath | six hours

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Prestridge, MD, Principal Investigator — Father Flanagan's Boys' Home; Sharad Kunnath, MD, Principal Investigator — Father Flanagan's Boys' Home
Locations (1):
- Boys Town National Research Hospital, Omaha, Nebraska, United States